CLINICAL TRIAL: NCT00418340
Title: Bacteria and Cytokines as Factors Modulating Visceral Afferent Processing in Irritable Bowel Syndrome: Manipulation of Intestinal Bacteria and Mucosal Cytokines by Probiotic Therapy and the Effect on Visceral Hypersensitivity
Brief Title: Manipulation of Visceral Sensitivity and Immune System in IBS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07.IBS.1
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome,; Visceral hypersensitivity,; probiotic therapy,; immune response
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics; Dietary Supplements

INTERVENTIONS:
Drug: probiotic (bacterial/dietary supplement)

SUMMARY:
Irritable bowel syndrome (IBS) is a common condition. At least 20% of the population suffer from IBS. The symptoms of abdominal pain, diarrhoea, constipation, bloating and difficulty with bowel motions are often disabling. Many of those affected are young and report a poor quality of life (QOL) to a degree that is similar to gut inflammatory conditions like ulcerative colitis and Crohn's disease. Yet the impact of IBS on patients' lives is often underestimated. This is probably because unlike inflammatory bowel disease, in which the bowel is inflammed and bleeds, the bowel in IBS looks normal. Instead the problem is of abnormal functioning of the gut the cause of which is unknown.

Currently therapy for IBS is limited and until recently therapy has focused on treating the symptoms to improve QOL primarily because the underlying mechanism of IBS is poorly understood. However as more processes are being implicated in IBS e.g. visceral hypersensitivity (excessive response to sensory stimuli within the gut), infection, immune activation, dysmotility and abnormal gut fermentation , the potential for new therapies looks promising. The evidence that gut bacteria play a role in inducing IBS symptoms is due to observations of an improvement of IBS symptoms with probiotic therapy (bacterial supplements) and antibiotic therapy.

Patients with IBS are hypersensitive to colorectal distension compared with healthy controls. Studies carried out in our unit have shown that visceral pain thresholds in response to stress are lower in patients with IBS compared with healthy volunteers. This hypersensitivity is apparent in response to both a physical and chemical stimulus but the triggers to visceral hypersensitivity remain largely unknown. Animal models suggest roles for both host immune response and intestinal bacteria in the induction of visceral hypersensitivity. This proposal will focus on further exploration of the mechanisms underlying visceral hypersensitivity to direct future targeting of therapy.

Previous independent studies showed that (a) bacteria reduce visceral hypersensitivity, (b)probiotic therapy can alter gut immune response and (c) gut sensation is affected by the type of immune cells in the gut. Our research proposal will investigate the relationship between gut bacteria, the immune system and the sensory gut nerves in order to understand how IBS symptoms are generated. This understanding will be the critical for effective future drug treatment.

DETAILED DESCRIPTION:
This research will study

1) probiotic-induced changes in visceral hypersensitivity and immune activity The effects of probiotic therapy will be assessed in a randomised placebo-controlled study. Subjects will be recruited prospectively from outpatient clinics. A flow chart of the study is shown in appendix 1 of the protocol. Patient selection. IBS patients will be selected according to inclusion and exclusion criteria.

Disease severity will be determined at enrolment with a validated IBS symptom questionnaire.

Questionnaires to exclude psychiatric illness: The well-validated Hospital Anxiety Depression Score (HADS)questionniaire will be used to identify patients with anxiety and depression. A SCL-90 questionnaire will also be used to assess the psychological profile of patients as this may have an impact on the response to therapy.

Probiotic therapy. Patients will be randomised to receive either VSL#3 (450 billion lyophilized bacteria/sachet) twice daily for 4 weeks or a placebo powder containing starch but no bacteria. VSL#3 was selected for use in this study because (a) it contains three different Bifidobacteria strains (in addition to lactobaccilli and streptococci) and the limited evidence available Bifidobacteria as the most effective probiotics in IBS 10; (b)it induces IL-10 production by intestinal DC 27 and, in pouchitis studies, stimulated IL-10 production in vivo 38; IBS has been associated with a deficiency in IL-10 production; (c) studies from one group have yielded promising results with this particular probiotic preparation.

1. Assessing the clinical response to therapy

   * Physiological response to probiotic therapy: Rectal sensitivity will be assessed at baseline and at day 28 of therapy. Rectal sensitivity to pressure and pain will be assessed with Barostat device and electrical stimulation respectively. Barostat device has been used in many other studies as a measure of sensation to pressure. Electrical stimulation is currently used in clinical practice. Equipment for both tests is currently in use at out physiology laboratory.
   * Symptomatic response to probiotic therapy: IBS symptom scores will be made at baseline and at d28 of therapy. The three symptoms of IBS will be assessed to determine response to therapy: abdominal pain/discomfort, bloating/ distension and bowel movements, each scored on an ordinal scale (Likert scale; maximum score 7) and on a 100mm visual analogue scale (VAS; maximum score 100). A composite score with the sums of the 3 cardinal symptoms will also be calculated for each patient (Likert scale maximum score 21) (VAS; maximum score 300).
   * Quality of life (QOL) with probiotic therapy: The SF-36 Heath-related QOL questionnaire, and the IBS QOL questionnaire will be administered at baseline and at day 28. This will assess the impact of IBS symptoms on the QOL and any changes following probiotic therapy. Follow-up: Patients will be contacted at 6 months to reassess symptom scores and QOL and determine longer-term impact of therapy.
2. Assessing Immunological response to probiotic therapy. Venepuncture will be performed for collection of blood immune cells at baseline and day 28. Colonic biopsies will be collected via a flexible sigmoidoscopy at entry baseline and at day 28 following the physiological tests. The biopsies will be use for analysis of cytokine production and to a limited phenotypic analysis of colonic immune cells (DC) with markers to be selected on the basis of data from an on-going cross-sectional study looking at DC in IBS compared to controls. Full analysis of blood DC will be performed at each time point. Changes in DC populations and cytokine production will be secondary endpoints of the study.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilling the Rome II criteria for the diagnosis of IBS
* normal blood investigations
* normal colonoscopy

Exclusion Criteria:

* a history of weight loss
* rectal bleeding
* fevers
* psychiatric illness (severe depression, anxiety, mania and schizophrenia)
* active infection
* recent antibiotic therapy or anti-inflammatory medication within previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-12

PRIMARY OUTCOMES:
The primary outcome measure is the change in physiological rectal sensitivity and before and after probiotic
therapy.

SECONDARY OUTCOMES:
Secondary outcome measures are the change symptoms and QOL induced by probiotic therapy and the
change in the immune response after probiotic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Naila Arebi, MD, PhD, MRCP, Principal Investigator — London North West Healthcare NHS Trust
Locations (1):
- North West London Hospitals NHS Trust - St Mark's, London, Middlesex, United Kingdom